CLINICAL TRIAL: NCT04312204
Title: Exploratory Clinical Trial of Sintilimab Combined With Gemcitabine/Carboplatin Regimen in the Treatment of Advanced Primary Pulmonary Lymphoepithelioma-like Carcinoma（LELC）
Brief Title: Clinical Trial of Sintilimab Combined With Gemcitabine/Carboplatin Regimen in the Treatment of Advanced Primary Pulmonary Lymphoepithelioma-like Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhou Chengzhi (Other)
Responsible Party: Sponsor-Investigator, Zhou Chengzhi, Professor, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CROC2001
Record Dates: First submitted 2020-03-12; First posted 2020-03-18 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Primary Pulmonary Lymphoepithelioma-like Carcinoma; Lung Cancer
Keywords: sintilimab; gemcitabine; Carboplatin; lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab+Gemcitabine+Carboplatin (Experimental)
  Interventions: Drug: Sintilimab combined with Gemcitabine and Carboplatin

INTERVENTIONS:
Drug: Sintilimab combined with Gemcitabine and Carboplatin — The patients will received Gemcitabine1000mg/m2(d1,d8)(iv)+carboplatin AUC 5 (d1)(iv),4 cycles, Sintilimab 200 mg (3mg/kg when the weight <40kg ) (d1) (iv) in one cycle every 3 weeks, until PD or death.
  Radiological examinations (according to the RECIST 1.1 criteria) at baseline will be repeated for tumor response evaluation following every two cycles of chemotherapy. Patients will be followed up to 30 days after the last dose of study chemotherapy, and then every 3 months.

SUMMARY:
The trial was designed to explore the safety and efficacy of sintilimab combined with gemcitabine and carboplatin in the treatment of advanced LELC.

ELIGIBILITY:
Inclusion Criteria:

* 1. age 18-75, male or female;
* 2. patients with advanced (inoperable stage iiiib -IV) primary pulmonary lymphoepithelioid carcinoma diagnosed pathologically, with at least one measurable lesion meeting RECIST v1.1 criteria;
* 3. patients have not received systemic therapy before (patients who have received platinum-containing adjuvant chemotherapy, neoadjuvant chemotherapy or radical chemoradiotherapy for advanced disease can enter if the disease progression occurs 6 months after the end of the last treatment);
* 4. ECOG PS: 0-1; expected survival ≥12 weeks;
* 5. vital organ functions meet the following requirements (excluding the use of any blood components or cytokines during screening) :The absolute count of neutrophils ≥1.5×109/L;Platelet ≥90×109/L;Hemoglobin ≥9g/dL;Serum albumin ≥3g/dL;Thyroid stimulating hormone (TSH) ≤ULN (if abnormal, T3 and T4 levels should be examined at the same time; if T3 and T4 levels are normal, they can be included in the group);Bilirubin ≤ULN;ALT and AST≤1.5 ULN;AKP 2.5 x ULN or less;Serum creatinine ≤1.5 ULN or creatinine clearance ≥60mL/min;
* 6. women of childbearing age must have been using reliable contraception or have had a pregnancy test (serum or urine) within 7 days prior to enrollment and have had negative results and be willing to use appropriate methods of contraception during the trial and 8 weeks after the last administration of the trial drug. For men, consent must be given to appropriate methods of contraception or surgical sterilization during the trial and 8 weeks after the last administration of the trial drug;
* 7. subjects voluntarily participate in this study and sign informed consent, with good compliance and follow up.

Exclusion Criteria:

* 1. those who have used other drugs to study drugs in clinical trials within 4 weeks before the first drug use;
* 2. the presence of any active autoimmune diseases or a history of autoimmune diseases (as follows, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, or decreased thyroid function; Subjects with vitiligo or with complete remission of asthma in childhood were included without any intervention in adulthood. Subjects with asthma requiring medical intervention with bronchodilators were not included.
* 3. subjects who are using immunosuppressive agents, or systemic, or absorbable local hormone therapy for immunosuppressive purposes (dose >10mg/ day prednisone or other therapeutic hormones) and continue to use within 2 weeks prior to enrollment;
* 4. severe allergic reaction to monoclonal antibody;
* 5. subjects with clinically symptomatic CNS metastases (e.g. cerebral edema, need for hormone intervention, or progression of brain metastases). Patients who have received previous treatment for brain or meningeal metastasis, such as clinical stability (MRI) has been maintained for at least 2 months, and who have stopped systemic sex hormone therapy (dose >10mg/ day prednisone or other therapeutic hormones) for more than 2 weeks can be included.
* 6. subjects have heart clinical symptoms or diseases that are not well controlled, such as: a. NYHA grade 2 or above heart failure; B. unstable angina pectoris; C. Had myocardial infarction within 1 year; D. Supraventricular or ventricular arrhythmias of clinical significance require treatment or intervention;
* 7. subjects who have previously received radiotherapy, chemotherapy, hormone therapy, surgery or molecular targeted therapy, and who have received less than 4 weeks before the study (or 5 drug half-lives, with the selected time) after the completion of the treatment (the last medication); Adverse events caused by previous treatment (except hair loss) did not recover to ≤ 1 degree CTCAE;
* 8. subjects with congenital or acquired immune deficiency (such as HIV infection) or active hepatitis (hepatitis b reference: HBsAg positive, HBV DNA≥2000 IU/ml or copy number ≥104/ml; Hepatitis c reference: positive HCV antibody;
* 9. subjects with active infection or unexplained fever >38.5 degrees during screening or before first administration;
* 10. subjects with congenital or acquired immune deficiency (such as HIV infection) or active hepatitis (hepatitis b reference: HBsAg positive, HBV DNA≥2000 IU/ml or copy number ≥104/ml; Hepatitis c reference: positive HCV antibody;
* 11. other malignancies (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix of the cervix) that the subjects had had or had at the same time;
* 12. according to the researcher's judgment, the subjects have other factors that may lead to the forced termination of this study, such as other serious diseases (including mental diseases) requiring combined treatment, severe laboratory examination abnormalities, accompanied by family or social factors, which may affect the safety of the subjects, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | Approximately 18 months
  ORR was defined as the percentage of participants with confirmed objective tumor response, complete response (CR) or partial response (PR), as determined by investigator using RECIST v1.1 criteria
safety(Adverse Events) | From the day the patient signs informed consent form until 30 days after last dose of sintilimab
  Safety will be assessed according to common terminology criteria for adverse events version 4.0 (CTC AE 4.0)
quality of life（the patient report outcome） | From the day the patient received treatment until 30 days after last dose of sintilimab
  Each patient answers to specific questions in questionnaire The time frame of most questions is "How would you rate your quality fo life during the last month"

CONTACTS AND LOCATIONS:
Locations (1):
- Zhou Chengzhi, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin X, Deng H, Fang N, Chen L, Chen R, Xie X, Xie Z, Zhang J, Liu M, Liu L, Sun N, Wang F, Yang Y, Lv X, Zhang Z, Cai S, Hou T, Li S, He J, Zhou C. Sintilimab plus chemotherapy for first-line treatment of advanced pulmonary lymphoepithelioma-like carcinoma: Phase 2 trial. Cell Rep Med. 2025 Oct 21;6(10):102398. doi: 10.1016/j.xcrm.2025.102398. Epub 2025 Oct 6. PMID 41056950